CLINICAL TRIAL: NCT04985266
Title: A Randomised Trial of Early Detection of Molecular Relapse With Circulating Tumour DNA Tracking and Treatment With Palbociclib Plus Fulvestrant Versus Standard Endocrine Therapy in Patients With ER Positive HER2 Negative Breast Cancer
Brief Title: A Trial of Early Detection of Molecular Relapse With Circulating Tumour DNA Tracking and Treatment With Palbociclib Plus Fulvestrant Versus Standard Endocrine Therapy in Patients With ER Positive HER2 Negative Breast Cancer
Acronym: TRAK-ER
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Collaborators: Pfizer (Industry); AstraZeneca (Industry); Institute of Cancer Research, United Kingdom (Other); UNICANCER (Other); Gustave Roussy, Cancer Campus, Grand Paris (Other); Invitae Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCR5316
Record Dates: First submitted 2021-06-25; First posted 2021-08-02 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: ER+ Breast Cancer; HER2-negative Breast Cancer
MeSH Terms: interventions — palbociclib; Fulvestrant; Tamoxifen; Letrozole; exemestane; Anastrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard endocrine therapy (Active Comparator): Standard endocrine therapy will continue for up to 24 months on trial.
  Standard endocrine therapies include tamoxifen, and aromatase inhibitors (letrozole, anastrazole, exemestane).
  Interventions: Drug: Tamoxifen; Drug: Letrozole; Drug: Exemestane; Drug: Anastrozole
- Palbociclib and fulvestrant (Experimental): Treatment with palbociclib plus fulvestrant will continue for a maximum of 24 months.
  Palbociclib will be given orally once a day on days 1-21 of each 28 day cycle.
  Fulvestrant 500 mg will be administered on cycle 1 days 1 and 15, cycle 2 day 1 and then every 28 days thereafter (plus or minus 3 days) as two intramuscular injections of 250mg fulvestrant at each visit.
  Interventions: Drug: Palbociclib 125Mg Tab; Drug: Fulvestrant injection

INTERVENTIONS:
Drug: Palbociclib 125Mg Tab — Palbociclib Tablets, 125 mg orally once daily, beginning on Cycle 1, on Days 1-21 of each 28-day cycle.
  Arms: Palbociclib and fulvestrant
Drug: Fulvestrant injection — Fulvestrant Intramuscular injections, 500 mg as two injection of 250mg fulvestrant in 5ml solution at each visit. No fulvestrant dose reductions are permitted. Administered on days 1, 15 (plus or minus 3 days), 29 (plus or minus 3 days), and every 28 (plus or minus 3 days) days thereafter.
  Arms: Palbociclib and fulvestrant
Drug: Tamoxifen — As per clinical guidelines
  Arms: Standard endocrine therapy
Drug: Letrozole — As per clinical guidelines
  Arms: Standard endocrine therapy
Drug: Exemestane — As per clinical guidelines
  Arms: Standard endocrine therapy
Drug: Anastrozole — As per clinical guidelines
  Arms: Standard endocrine therapy

SUMMARY:
Detection of molecular relapse with circulating tumour DNA analysis can identify which patients with ER positive breast cancer are relapsing on adjuvant endocrine therapy. This trial will aim to demonstrate that palbociclib and fulvestrant, can defer or prevent relapse in patients with ctDNA detected molecular relapse.

The TRAK-ER trial will have two phases, a ctDNA surveillance phase and a randomised therapy trial in patients with positive ctDNA.

The TRAK-ER trial will establish a ctDNA screening programme for patients with ER positive breast cancer receiving adjuvant endocrine therapy with at least a further three years of standard adjuvant endocrine therapy planned. Patients recruited into the TRAK-ER study will have high-risk clinical features to identify patients at higher risk of future relapse.

ctDNA assays will be used to identify which people are at very high risk of relapse (i.e. those with a positive ctDNA result), and randomise this high risk population between standard endocrine therapy versus palbociclib plus fulvestrant for up to two years.

DETAILED DESCRIPTION:
The TRAK-ER trial is a multi-centre, randomised, open-label trial in patients with early stage oestrogen reception positive (ER+) human epidermal growth receptor-2 negative (HER2-) breast cancer, whom have detectable circulating DNA (ctDNA) but no overt macroscopic disease on imaging. TRAK-ER aims to demonstrate that fulvestrant plus palbociclib improves relapse free survival compared to standard endocrine therapy in this patient group.

Despite current treatment, patients with ER+HER2- breast cancer are considered high-risk of distant recurrence for more than the first two decades after initial diagnosis. ctDNA analysis provides a non-invasive, serial source of tumour material which can monitor tumour dynamics and detect molecular relapse.

TRAK-ER will be split into two phases, the first surveillance phase aims to investigate the use of ctDNA to identify and predict the risk of molecular relapse in early ER+/HER2- breast cancer patients whom are receiving adjuvant endocrine therapy with no overt macroscopic disease on imaging. Using ctDNA assays, patients enrolled on TRAK-ER will receive ctDNA testing on a three-monthly basis for up to three years. In the instance where ctDNA is detected, imaging will determine whether overt disease is present. If a patient had a positive ctDNA detection and no macroscopic disease on the staging scan, the patient will be randomised to one of the treatment groups in the second phase of TRAK-ER, the treatment phase.

The treatment phase of TRAK-ER will be a randomised, open-label study which aims to determine whether fulvestrant plus palbociclib (intervention arm) improves relapse free survival compared to standard endocrine therapy (control arm) in patients carried through from the surveillance phase. Patients on each arm will receive treatment (fulvestrant plus palbociclib or standard endocrine therapy) for up to 24 months. Six monthly imaging will determine the presence of macroscopic disease. If macroscopic disease is observed, the patient will discontinue TRAK-ER treatment and commence standard therapy outside of the TRAK-ER trial.

ELIGIBILITY:
Inclusion Criteria for ctDNA Surveillance:

1. Written informed consent to participate in the trial and to donation of tissue and blood samples
2. Male or female patients aged 18 years or older
3. ECOG performance status 0, 1 or 2 (see https://ecog-acrin.org/resources/ecog-performance-status)
4. Histologically proven primary ER+ (Allred score 6/8 or greater, or stain in ≥10% of cancer cells) and HER2- (immunohistochemistry 0/1+ and/or negative by in situ hybridization) breast cancer as determined by local laboratory
5. Patients with high risk early stage breast cancer according to at least one of the following criteria:

   Primary surgery (no other treatment prior to surgery) A. Four or more involved axillary lymph nodes or positive supraclavicular lymph node at diagnosis, or

   B. Tumour size > 5 cm, regardless of lymph node status, or

   C. 1-3 involved axillary lymph nodes and at least one of the following; i) Tumour size > 3 cm, ii) histological grade 3 iii) high genomic risk defined as Oncotype Dx Recurrence Score >=26, Prosigna score >=60, EPclin risk score >=4.0, or Mammaprint high risk category, or

   Neoadjuvant chemotherapy (chemotherapy prior to surgery)

   D. At least one lymph node positive (micrometastasis or macrometastasis) after chemotherapy

   E. Lymph node negative and tumour size > 3 cm after chemotherapy

   Neoadjuvant endocrine therapy (endocrine based therapy prior to surgery) Use the primary surgery criteria - staging tumour size and lymph node status may be either the pathological staging after endocrine therapy or on the initial clinical staging prior to neoadjuvant therapy
6. Available tissue from one archival tumour tissue sample (either from diagnostic biopsy, primary surgery or where available residual disease post-neoadjuvant chemotherapy)
7. No evidence of macroscopic distant metastatic disease or incurable locally advanced disease on staging scans conducted at any time since initial diagnosis.
8. Patients receiving standard endocrine therapy with aromatase inhibitors (letrozole, anastrazole, exemestane), tamoxifen, or combination of such for a minimum of 6 months* and maximum of 7 years duration with an additional three years of endocrine therapy planned. Pre- or peri-menopausal patients may also receive GnRH analogues.

   * patients may enrol during the first 6 months of standard endocrine therapy, and wait until at least 6 months of endocrine therapy has been received prior to starting ctDNA surveillance
9. Patients must have had surgery achieving clear margins (as per local guidelines)
10. Female and male patients of reproductive potential must be willing to use an adequate method of contraception for the first three years of the trial, if randomised to standard endocrine therapy for the duration of trial treatment through to at least 4 weeks after the last dose of trial treatment, and if randomised to fulvestrant and palbociclib to 2 years after the last dose of fulvestrant (see section 4.6). Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient.
11. Patients willing to have frequent blood tests.

Inclusion Criteria for Interventional phase:

1. Signed informed consent for treatment
2. ECOG performance status 0, 1 or 2
3. Women of childbearing potential should have a negative serum pregnancy test prior to randomisation. If randomisation occurs more than 72 hours prior to receiving the first dose of treatment the test must be repeated before treatment.
4. Female and male patients of childbearing potential must be willing to use an adequate method of contraception (section 4.6), starting with the first dose of treatment through 4 weeks after the last dose of treatment if randomised to standard endocrine therapy and 2 years after the last dose of fulvestrant if randomised to fulvestrant and palbociclib. Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the patient. Female patients will be deemed not of childbearing potential if they are postmenopausal or have had irreversible sterilisation
5. Patient has adequate bone marrow and organ function as defined by the following laboratory values:

   1. Absolute Neutrophil Count (ANC) ≥ 1.5 × 109/L
   2. Platelets ≥ 100 × 109/L
   3. Haemoglobin ≥ 100 g/L
   4. INR ≤1.5
   5. Creatinine <1.5 x ULN and creatinine clearance ≥30ml/min
   6. Total bilirubin < ULN except for patients with Gilbert's syndrome who may only be included if the total bilirubin is ≤ 3.0 × ULN or direct bilirubin ≤ 1.5 × ULN.
   7. Alanine aminotransferase (ALT) < 2.5 x ULN
   8. Aspartate aminotransferase (AST) < 2.5 × ULN
6. Patients must be post-menopausal OR

Pre- or peri-menopausal patients or men may be enrolled if they have ovarian/gonadal suppression with licensed GnRH analogues. Patients must have commenced licensed GnRH analogues at least 2 weeks prior to Cycle 1 Day 1 and continue throughout the study if randomised to fulvestrant and palbociclib.

Post-menopausal female patients, as defined by at least one of the following:

* Age ≥60 years;
* Age <60 years and cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause, and serum estradiol and FSH levels within the institutional laboratory's reference range for post-menopausal females;
* Documented bilateral oophorectomy;

Exclusion Criteria for ctDNA Surveillance:

1. Any concurrent or planned treatment for the current diagnosis of breast cancer other than adjuvant endocrine therapy or a bisphosphonate.
2. Patients with prior exposure to a CDK 4/6 inhibitor as part of standard of care may enrol only after at least 12 months from completing CDK4/6 therapy.
3. Prior exposure to therapeutic dose of fulvestrant is not permitted. One subtherapeutic dose of fulvestrant is permitted.
4. Prior diagnosis of cancer including prior diagnosis of breast cancer in the previous 5 years, other than for non-melanoma carcinoma of the skin or cervical carcinoma in situ
5. Patients previously entered into a therapeutic trial where experimental therapy is continued post-surgery. Patients who have entered a clinical trial of a CDK4/6 inhibitor in the adjuvant setting are not eligible. Patients who received a CDK4/6 inhibitor only before an operation, with no post-operative adjuvant use, are eligible.
6. Treatment with an unlicensed or investigational product within 4 weeks prior registration to trial
7. Patient has not recovered to ≤ grade 1 (except alopecia or certain other toxicities, which in the opinion of the Investigator should not exclude the patient) from related side effects of any prior antineoplastic therapy, not including side-effects of endocrine therapy
8. Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral medication (e.g. Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection)
9. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator' opinion cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol.
10. Clinically significant uncontrolled heart disease including any of the following:

    1. History of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to trial entry
    2. Symptomatic congestive heart failure
    3. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
    4. Cardiac arrhythmia.
11. History of pneumonitis, interstitial lung disease or pulmonary fibrosis
12. Known history of Human Immunodeficiency Virus (HIV) (testing not required as part of study screening)
13. Known active Hepatitis B or Hepatitis C (testing not required as part of study screening)
14. Females who are known to be pregnant or breastfeeding
15. History of bleeding diathesis (i.e. disseminated intravascular coagulation, clotting factor deficiency), other known abnormalities in coagulation or treatment with anticoagulants. Low molecular weight heparin (LMWH), low dose aspirin or clopidogrel are permitted.
16. Child-Pugh class C hepatic impairment or creatinine clearance < 30ml/min.
17. Patient with bilateral tumours, or unilateral multifocal cancers with multiple separate primary cancers.(Multifocal cancer that reflects a single primary cancer, in the opinion of the investigator, are eligible)

Exclusion Criteria for Interventional phase:

1. Evidence of recurrent disease (metastatic or local, see section 6.6 for management of patients with potentially curable local recurrences) on staging scans conducted since positive ctDNA result
2. Known hypersensitivity to the excipients of palbociclib plus fulvestrant
3. Any anti-cancer treatment since enrolling in the TRAK-ER study other than hormonal therapy or a bisphosphonate. Prior exposure to fulvestrant is not permitted.
4. Diagnosis of an alternative cancer since enrolment in the trial other than non-melanoma cancer of the skin or cervical carcinoma in situ
5. Patient has had major surgery within 4 weeks prior to starting trial treatment or has not recovered from major side effects of such procedure
6. Patient is currently receiving warfarin or other coumarin derived anti-coagulant, for treatment, prophylaxis or otherwise. Therapy with unfractionated heparin, low molecular weight heparin (LMWH), or a direct-acting oral anticoagulant (DOAC such as rivaroxaban or fondaparinux) is allowed
7. Patient has not recovered to ≤ grade 1 (except alopecia or certain other toxicities, which in the opinion of the Investigator should not exclude the patient) from related side effects of any prior antineoplastic therapy, not including side-effects of endocrine therapy
8. Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of oral medication (e.g. Crohn's disease, ulcerative diseases, uncontrolled nausea, vomiting, diarrhoea, malabsorption syndrome, or small bowel resection)
9. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the Investigator' opinion cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol.
10. Clinically significant uncontrolled heart disease including any of the following:

    1. History of myocardial infarction (MI), angina pectoris, symptomatic pericarditis, or coronary artery bypass graft (CABG) within 6 months prior to trial entry
    2. Symptomatic congestive heart failure
    3. Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome.
    4. Cardiac arrhythmia.
11. Patient is currently receiving any of the following substances and cannot be discontinued 7 days prior to Cycle 1 Day 1:

    * Medications that are strong inducers or inhibitors of CYP3A4 (section 8.5.2)
    * Herbal preparations/medications, dietary supplements, fruits (e.g grapefruit, pomelos, starfruit, Seville oranges) and their juice
12. History of pneumonitis, interstitial lung disease or pulmonary fibrosis
13. Known history of HIV (testing not required as part of study screening)
14. Known active Hepatitis B or Hepatitis C (testing not required as part of study screening)
15. Patient has a history of non-compliance to medical regimen
16. History of bleeding diathesis (i.e. disseminated intravascular coagulation, clotting factor deficiency), other known abnormalities in coagulation or treatment with anticoagulants. Low molecular weight heparin (LMWH), low dose aspirin or clopidogrel are permitted.
17. Females who are known to be pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1100 (Estimated)
Dates: Start 2022-03-30 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2030-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of positive ctDNA result during surveillance (Surveillance phase) | Up to 36 months from entry to study
  Test during the surveillance phase detects presence of ctDNA
Incidence of positive ctDNA result at first test (Surveillance phase) | Start of study
  Test during the surveillance phase detects presence of ctDNA in the first test
Relapse free survival (Treatment phase) | 60 months from randomisation
  Time from randomization to invasive local/regional recurrence (including ipsilateral invasive breast recurrence) or distant recurrence or death from any cause. Patients with second primary invasive cancers (breast or non-breast) would be censored at time of detection.

SECONDARY OUTCOMES:
Frequency and Severity of adverse events | up to 24 months from randomisation
  Frequency and severity of Adverse Events (AEs) assessed as per CTCAE v5
Overall survival | up to 60 months from randomisation
  Time from randomisation to death from any cause
Invasive disease free survival | up to 60 months from randomisation
  Time from randomisation to invasive local/regional recurrence (including ipsilateral invasive breast recurrence), new breast cancer (ipsilateral or contralateral) or distant recurrence or death from any cause. Patients with non-invasive recurrences or second primary invasive cancers (non-breast) would be censored at time of detection.
Distant recurrence free survival | up to 60 months from randomisation
  Time from randomization to distant invasive breast cancer recurrence or death from any cause. Patients with new contralateral invasive breast cancers or second primary invasive non-breast cancers would be censored at time of detection.
EQ-5D-5L quality of life assessment: Mobility element | up to 24 months from randomisation
  Assessed using the 5-point scale.
EQ-5D-5L quality of life assessment: Self-care element | up to 24 months from randomisation
  Assessed using the 5-point scale.
EQ-5D-5L quality of life assessment: Usual activities element | up to 24 months from randomisation
  Assessed using the 5-point scale.
EQ-5D-5L quality of life assessment: Pain/ Discomfort element | up to 24 months from randomisation
  Assessed using the 5-point scale.
EQ-5D-5L quality of life assessment: Anxiety/ Depression element | up to 24 months from randomisation
  Assessed using the 5-point scale.
EQ-5D-5L quality of life assessment: Visual Analogue Scale | up to 24 months from randomisation
  Assessed using 0-100 scale.

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Turner, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (49):
- France (21):
  - Institut de Cancérologie de l'Ouest, Angers
  - Centre Hospitalier Annecy Genevois_Site d'Annecy, Annecy
  - Institut du Cancer Avignon Sainte Catherine, Avignon
  - Centre Hospitalier Simone Veil de Blois, Blois
  - Institut Bergonié, Bordeaux
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre George François Leclerc, Dijon
  - Groupe Hospitalier Mutualiste de Grenoble, Grenoble
  - Clinique Chénieux, Limoges
  - Centre Hospitalier Universitaire de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancérologie de l'Ouest, Nantes
  - Centre Antoine Lacassagne, Nice
  - Gustave Roussy Cancer Campus, Paris
  - Hôpital Américain de Paris, Paris
  - Institut Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - CHU de Saint Etienne-Institut de Cancérologie, Saint-Priest-en-Jarez
  - Institut Claudius Regaud, Toulouse
- United Kingdom (28):
  - Barnet Hospital, London, Barnet
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - University Hospitals Dorset: Royal Bournemouth Hospital, Bournemouth
  - Royal Sussex Hospital, Brighton
  - Bristol Haematology and Oncology Centre, Bristol
  - Velindre Cancer Centre, Cardiff
  - Velindre University NHS Trust, Cardiff
  - Darlington Memorial Hospital, Darlington
  - Western General, Edinburgh
  - Royal Devon and Exeter Hospital, Exeter
  - Beatson West of Scotland Cancer Centre, Glasgow
  - North West Anglia NHS Foundation Trust: Hinchingbrooke Hospital, Huntingdon
  - St James's University Hospital, Leeds
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Liverpool
  - Barts Health NHS Trust, London
  - Mount Vernon Hospital, London
  - University College London Hospital, London
  - The Royal Free Hospital, London
  - The Royal Marsden NHS Foundation Trust, London
  - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hopsitals NHS Trust, Nottingham
  - Oxford Cancer & Haematology Centre, Churchill Hospital,, Oxford
  - North West Anglia NHS Foundation Trust: Peterborough Hospital, Peterborough
  - Derriford Hospital - UHPNT, Plymouth
  - University Hospitals Dorset: Poole Hospital, Poole
  - Weston Park Hospital, Sheffield
  - Somerset NHS Foundation Trust, Taunton

REFERENCES:
- [Background] Dawson SJ, Tsui DW, Murtaza M, Biggs H, Rueda OM, Chin SF, Dunning MJ, Gale D, Forshew T, Mahler-Araujo B, Rajan S, Humphray S, Becq J, Halsall D, Wallis M, Bentley D, Caldas C, Rosenfeld N. Analysis of circulating tumor DNA to monitor metastatic breast cancer. N Engl J Med. 2013 Mar 28;368(13):1199-209. doi: 10.1056/NEJMoa1213261. Epub 2013 Mar 13. PMID 23484797
- [Background] O'Leary B, Cutts RJ, Liu Y, Hrebien S, Huang X, Fenwick K, Andre F, Loibl S, Loi S, Garcia-Murillas I, Cristofanilli M, Huang Bartlett C, Turner NC. The Genetic Landscape and Clonal Evolution of Breast Cancer Resistance to Palbociclib plus Fulvestrant in the PALOMA-3 Trial. Cancer Discov. 2018 Nov;8(11):1390-1403. doi: 10.1158/2159-8290.CD-18-0264. Epub 2018 Sep 11. PMID 30206110
- [Background] Abbosh C, Birkbak NJ, Wilson GA, Jamal-Hanjani M, Constantin T, Salari R, Le Quesne J, Moore DA, Veeriah S, Rosenthal R, Marafioti T, Kirkizlar E, Watkins TBK, McGranahan N, Ward S, Martinson L, Riley J, Fraioli F, Al Bakir M, Gronroos E, Zambrana F, Endozo R, Bi WL, Fennessy FM, Sponer N, Johnson D, Laycock J, Shafi S, Czyzewska-Khan J, Rowan A, Chambers T, Matthews N, Turajlic S, Hiley C, Lee SM, Forster MD, Ahmad T, Falzon M, Borg E, Lawrence D, Hayward M, Kolvekar S, Panagiotopoulos N, Janes SM, Thakrar R, Ahmed A, Blackhall F, Summers Y, Hafez D, Naik A, Ganguly A, Kareht S, Shah R, Joseph L, Marie Quinn A, Crosbie PA, Naidu B, Middleton G, Langman G, Trotter S, Nicolson M, Remmen H, Kerr K, Chetty M, Gomersall L, Fennell DA, Nakas A, Rathinam S, Anand G, Khan S, Russell P, Ezhil V, Ismail B, Irvin-Sellers M, Prakash V, Lester JF, Kornaszewska M, Attanoos R, Adams H, Davies H, Oukrif D, Akarca AU, Hartley JA, Lowe HL, Lock S, Iles N, Bell H, Ngai Y, Elgar G, Szallasi Z, Schwarz RF, Herrero J, Stewart A, Quezada SA, Peggs KS, Van Loo P, Dive C, Lin CJ, Rabinowitz M, Aerts HJWL, Hackshaw A, Shaw JA, Zimmermann BG; TRACERx consortium; PEACE consortium; Swanton C. Phylogenetic ctDNA analysis depicts early-stage lung cancer evolution. Nature. 2017 Apr 26;545(7655):446-451. doi: 10.1038/nature22364. PMID 28445469
- [Background] Bettegowda C, Sausen M, Leary RJ, Kinde I, Wang Y, Agrawal N, Bartlett BR, Wang H, Luber B, Alani RM, Antonarakis ES, Azad NS, Bardelli A, Brem H, Cameron JL, Lee CC, Fecher LA, Gallia GL, Gibbs P, Le D, Giuntoli RL, Goggins M, Hogarty MD, Holdhoff M, Hong SM, Jiao Y, Juhl HH, Kim JJ, Siravegna G, Laheru DA, Lauricella C, Lim M, Lipson EJ, Marie SK, Netto GJ, Oliner KS, Olivi A, Olsson L, Riggins GJ, Sartore-Bianchi A, Schmidt K, Shih lM, Oba-Shinjo SM, Siena S, Theodorescu D, Tie J, Harkins TT, Veronese S, Wang TL, Weingart JD, Wolfgang CL, Wood LD, Xing D, Hruban RH, Wu J, Allen PJ, Schmidt CM, Choti MA, Velculescu VE, Kinzler KW, Vogelstein B, Papadopoulos N, Diaz LA Jr. Detection of circulating tumor DNA in early- and late-stage human malignancies. Sci Transl Med. 2014 Feb 19;6(224):224ra24. doi: 10.1126/scitranslmed.3007094. PMID 24553385
- [Background] Garcia-Murillas I, Chopra N, Comino-Mendez I, Beaney M, Tovey H, Cutts RJ, Swift C, Kriplani D, Afentakis M, Hrebien S, Walsh-Crestani G, Barry P, Johnston SRD, Ring A, Bliss J, Russell S, Evans A, Skene A, Wheatley D, Dowsett M, Smith IE, Turner NC. Assessment of Molecular Relapse Detection in Early-Stage Breast Cancer. JAMA Oncol. 2019 Oct 1;5(10):1473-1478. doi: 10.1001/jamaoncol.2019.1838. PMID 31369045
- [Background] Garcia-Murillas I, Schiavon G, Weigelt B, Ng C, Hrebien S, Cutts RJ, Cheang M, Osin P, Nerurkar A, Kozarewa I, Garrido JA, Dowsett M, Reis-Filho JS, Smith IE, Turner NC. Mutation tracking in circulating tumor DNA predicts relapse in early breast cancer. Sci Transl Med. 2015 Aug 26;7(302):302ra133. doi: 10.1126/scitranslmed.aab0021. PMID 26311728
- [Background] Turner NC, Ro J, Andre F, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Huang Bartlett C, Zhang K, Giorgetti C, Randolph S, Koehler M, Cristofanilli M; PALOMA3 Study Group. Palbociclib in Hormone-Receptor-Positive Advanced Breast Cancer. N Engl J Med. 2015 Jul 16;373(3):209-19. doi: 10.1056/NEJMoa1505270. Epub 2015 Jun 1. PMID 26030518
- [Background] Finn RS, Martin M, Rugo HS, Jones S, Im SA, Gelmon K, Harbeck N, Lipatov ON, Walshe JM, Moulder S, Gauthier E, Lu DR, Randolph S, Dieras V, Slamon DJ. Palbociclib and Letrozole in Advanced Breast Cancer. N Engl J Med. 2016 Nov 17;375(20):1925-1936. doi: 10.1056/NEJMoa1607303. PMID 27959613
- [Background] Turner NC, Slamon DJ, Ro J, Bondarenko I, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Loibl S, Andre F, Puyana Theall K, Huang X, Giorgetti C, Huang Bartlett C, Cristofanilli M. Overall Survival with Palbociclib and Fulvestrant in Advanced Breast Cancer. N Engl J Med. 2018 Nov 15;379(20):1926-1936. doi: 10.1056/NEJMoa1810527. Epub 2018 Oct 20. PMID 30345905
- [Background] Asghar U, Witkiewicz AK, Turner NC, Knudsen ES. The history and future of targeting cyclin-dependent kinases in cancer therapy. Nat Rev Drug Discov. 2015 Feb;14(2):130-46. doi: 10.1038/nrd4504. PMID 25633797
- [Background] Di Leo A, Jerusalem G, Petruzelka L, Torres R, Bondarenko IN, Khasanov R, Verhoeven D, Pedrini JL, Smirnova I, Lichinitser MR, Pendergrass K, Garnett S, Lindemann JP, Sapunar F, Martin M. Results of the CONFIRM phase III trial comparing fulvestrant 250 mg with fulvestrant 500 mg in postmenopausal women with estrogen receptor-positive advanced breast cancer. J Clin Oncol. 2010 Oct 20;28(30):4594-600. doi: 10.1200/JCO.2010.28.8415. Epub 2010 Sep 20. PMID 20855825
- [Background] Di Leo A, Jerusalem G, Petruzelka L, Torres R, Bondarenko IN, Khasanov R, Verhoeven D, Pedrini JL, Smirnova I, Lichinitser MR, Pendergrass K, Malorni L, Garnett S, Rukazenkov Y, Martin M. Final overall survival: fulvestrant 500 mg vs 250 mg in the randomized CONFIRM trial. J Natl Cancer Inst. 2014 Jan;106(1):djt337. doi: 10.1093/jnci/djt337. Epub 2013 Dec 7. PMID 24317176